CLINICAL TRIAL: NCT04993339
Title: Clinical Outcomes of ACL Reconstruction Augmented by an Injectable Osteoconductive/Osteoinductive Compound
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Francesco Travascio, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20150981
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Surgery (No Intervention): Participants in this group undergoing standard of care reparative surgery will not receive additional intervention
- Standard Surgery with OOC (Experimental): Participants in this group undergoing standard of care reparative surgery will receive OOC as an additional intervention
  Interventions: Drug: OOC

INTERVENTIONS:
Drug: OOC — The OOC will be mixed with autologous 5cc of platelet rich plasma (PRP), and then injected using a syringe into both tibia and femoral tunnels
  Other Names: StimuBlast
  Arms: Standard Surgery with OOC

SUMMARY:
The goal of this study is to determine whether the use of injectable osteoinductive/osteoconductive compounds (OOC) during Anterior Cruciate Ligament (ACL) reconstructive surgery, combined with an accelerated rehabilitation protocol (ARP) provides clinical outcomes superior to those attained via traditional ACL reconstruction and delayed rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* any adult undergoing a surgical procedure for hamstring ACL reconstruction

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Travascio, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Surgery | Standard Surgery With OOC
Started | 14 | 12
Completed | 11 | 10
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — no MRI scan | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Surgery | Standard Surgery With OOC | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bone Tunnel Expansion
Description: Number of participants will be classified with having femoral and tibial tunnel expansion as:
  * minimal expansion (<1mm)
  * mild expansion (<5mm)
  * moderate expansion (5-10mm)
  * large expansion (>10mm)
  as measured via Magnetic Resonance Imaging (MRI)
Time Frame: up to 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Surgery | Standard Surgery With OOC
Number analyzed (Participants) | 11 | 10
Participants
  femoral minimal expansion | 0 | 4
  femoral mild expansion | 10 | 6
  femoral moderate expansion | 1 | 0
  femoral large expansion | 0 | 0
  tibial minimal expansion | 0 | 3
  tibial mild expansion | 8 | 7
  tibial moderate expansion | 2 | 0
  tibial large expansion | 1 | 0

2. Secondary Outcome: Graft Maturation
Description: as measured in millimeters via Magnetic Resonance Imaging (MRI)
Time Frame: up to 12 months post-surgery
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Standard Surgery | Standard Surgery With OOC
Number analyzed (Participants) | 11 | 10
millimeters | 4.28 (2.55) | 2.28 (1.97)

3. Secondary Outcome: Number of Participants With Tunnel Ganglion Cyst Formation
Description: as measured via Magnetic Resonance Imaging (MRI)
Time Frame: up to 12 months post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Surgery | Standard Surgery With OOC
Number analyzed (Participants) | 11 | 10
Participants | 8 | 2

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Surgery | Standard Surgery With OOC
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT04993339/Prot_SAP_000.pdf